CLINICAL TRIAL: NCT06932276
Title: Effectiveness of an Evidence-based Intervention to Promote Smoke-free Homes: a Randomised Controlled Trial
Brief Title: Implementing an Adapted Smoke-free Homes Intervention in Spain
Acronym: SFH Spain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: Emory University (Other); Public Health Agency of Barcelona (Other); Agència de Salut Pública de Catalunya (ASPCAT) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHF-Spain; PI21/00818 (Other Grant/Funding Number: Instituto de Salud Carlos III (Spanish national grant))
Record Dates: First submitted 2025-04-01; First posted 2025-04-17 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Secondhand Tobacco Smoke Exposure Reduction; Smoking Prevention
Keywords: smoke-free homes; Spain

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial: randomization at level of Assotiation of Students Families (ASF, i.e. school). All participants from the same ASF will be either in the intervention or a control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants will receive an adapted version of the "Some Things Are Better Outside" intervention, designed to encourage them to voluntarily create a smoke-free home by accepting a norm of never smoking at home, whether indoors or outdoors, such as on balconies. The intervention is delivered over six weeks and consists of four components: an initial mailing of printed materials, a coaching call, and two additional mailings. It is based on five steps to adopting a smoke-free home: 1) deciding on the reasons for creating one, 2) discussing it with family members, 3) choosing a date to go smoke-free, 4) making the home a smoke-free environment, and 5) maintaining it as smoke-free.
  Interventions: Behavioral: "Some things a re better outside"
- Control (No Intervention): Participants in the intervention group will not receive the intervention. However, all participants in the control group will be offered the intervention after the final follow-up, which takes place six months post-baseline.

INTERVENTIONS:
Behavioral: "Some things a re better outside" — "Some Things Are Better Outside" interventionis designed to encourage participants to voluntarily create a smoke-free home by accepting a norm of never smoking at home, whether indoors or outdoors, such as on balconies. The intervention is delivered over six weeks and consists of four components: an initial mailing of printed materials, a coaching call, and two additional mailings. It is based on five steps to adopting a smoke-free home: 1) deciding on the reasons for creating one, 2) discussing it with family members, 3) choosing a date to go smoke-free, 4) making the home a smoke-free environment, and 5) maintaining it as smoke-free.
  Arms: Intervention

SUMMARY:
While smoking and exposure to second-hand tobacco smoke (SHS) in most public places is addressed by smoke-free regulations, the exposure to SHS at private places, such as homes, is still prevalent in Spain and represents a significant public health challenge.

Main objective of the study: to evaluate the effectiveness of an evidence-based intervention to create smoke-free homes in households with children.

Design: cluster randomised controlled trial. Target population: families with children (≤18 years old) and at least one smoker who allow smoking in the home.

Sample: 51 clusters per group (intervention and control) with an average 4 participants per cluster. In total, 102 schools and 408 participants.

Recruitment: The Tobacco Control Unit, the study promoter, will invite the Associations of the Students' Families (ASF) of schools in the Metropolitan Area of Barcelona to join the study. Those ASFs that participate, will run an information campaign among their members (caregivers of students enrolled at each school) explaining them the study and providing a link to sign up for it via a designated Website. Tobacco Control Unit Research Team will then contact the potential participants and start their participation.

The intervention is an adapted intervention "Some things a better outside" developed by the Emory University. The intervention is based on 5 steps (Decide; Talk; Pick a date; Make it happen; and Keep it up) and is delivered during 6 weeks in 2-week intervals (first mailing, counselling call, and two other mailings). The intervention will be delivered only to the IG participants in the CG will not receive the intervention but may optionally receive it following the 6 months follow-up.

Data collection: 1) baseline; 2) at month 3 postbaseline; 3) at month 6 postbaseline. Primary outcome: prevalence of households with complete smoking ban in the homes at follow-ups (self-reported). Secondary outcomes: SHS exposure level at follow-ups (self-reported).

DETAILED DESCRIPTION:
Second-hand tobacco smoke (SHS) is a mixture of smoke exhaled by a smoker and smoke from the burning end of a cigarette. There are more than 4,000 components in SHS, including toxic substances, irritants and, approximately 70 carcinogens. Since 2004, SHS is defined as carcinogenic to humans (Group 1) by the International Agency for Research on Cancer. Exposure to SHS is an important public health problem as it causes a number of life-threatening diseases, among others lung cancer, stroke, chronic obstructive pulmonary disease, and ischemic heart disease in adults. Moreover, children exposed to SHS are at an increased risk for sudden infant death syndrome, acute respiratory infections, otitis media, and more severe asthma. Globally, SHS exposure was the 13th-leading risk factor for deaths in 2019, accounting for 1.30 million deaths. It contributed to 37.0 million disability adjusted life years worldwide, with 11.2% of the burden seen among children under the age of 5 years. While exposure to SHS in most public places is addressed by smokefree regulations, smoking and, consequently, the exposure to SHS at private places, such as homes, is still prevalent and represents a significant public health challenge.

It is evaluated that globally approximately 40% of youth is exposed to SHS at home. In a survey conducted among schoolchildren in Terrassa (Barcelona) in 2006 we found similar results, 41% of children aged 12-13 years reported exposure to SHS at home. For younger ages, another survey we conducted in Barcelona in 2016 showed that 71% of children younger than 12 years were exposed to SHS and 26% of them were exposed to SHS at home. Previous research in Spain have shown that SHS exposure at home is strongly correlated with family structure, smoking rules in household, number of smokers and non-smokers at home and number of cigarettes smoked; moreover, social disparities exist in SHS exposure among children and therefore, the inequalities in SHS burden persist in the local population.

In Spain, a few initiatives have been undertaken to reduce SHS exposure in children. In 2006, the RESPIR·NET multi-level (individual, family, and school) school-based intervention to prevent the exposure to SHS among schoolchildren (12-14 years old) was developed and tested in the city of Terrassa (Barcelona). While crude data indicated that in the intervention group SHS exposure significantly decreased at home (-16.9%); after adjustment for potential confounders the changes showed to be non-significant. In 2008-2009, the BIBE study aimed to evaluate a brief intervention within the context of primary health care, directed to parents who smoke, in order to reduce SHS exposure of babies. A multicentre, open, cluster-randomised clinical trial showed that parents who received the intervention to avoid SHS better adopted the recommended strategies at home with reduced nicotine concentrations in babies' hair samples.

While these interventions did not target promotion of smoke-free homes specifically, a recent study, part of a larger TackSHS Project (www.tackshs.eu), aimed to design, implement and evaluate a "Measuring for change" intervention to create smoke-free homes among families with children from disadvantaged areas. The intervention, developed by the team of the University of Stirling, is based on providing remote air quality feedback to the participants via short messages and emails. While the intervention resulted in small but significant reduction of SHS exposure, it was not effective in creating smoke-free homes; in addition, the design requiring two home visits and installation of air quality monitors challenged the participants' recruitment.

In summary, currently in Spain a high proportion of households allow smoking resulting in unneglectable prevalence and burden of exposure to SHS at home among adults and children. No comprehensive and systematic support is offered at national or local levels for those who want to create smoke-free homes resulting in a significant gap in health prevention services. Therefore, there is an important need to offer such services to Spanish population.

The solution: adopting an evidence-based smoke-free intervention. In response to this need, we will test the effectiveness of an adapted brief evidence-based intervention to promote smoke-free homes initially developed by the University of Emory (PI: Prof. Michelle Kegler). This intervention was adopted, piloted and tested in a number of the US States and cities with excellent results, that given its minimal intervention nature, enables reaching a greater number of people. Additionally, the proposed intervention will target families with children to increase the potential impact on health burden from a reduced SHS exposure at homes. We aim to test the intervention in Catalonia with a view to its future scalability at the national level, ensuring comprehensive support for creating smoke-free homes as part of a service package available to schools and associations of students' families. Therefore, the main aim of this study is to evaluate the effectiveness of an evidence-based intervention to create smoke-free homes in households with children.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* Live in a household with at least one minor (younger than 18 years old)
* Live in a household with at least one person who smokes
* Smoking is allowed at home (always or sometimes; everywhere or in some specific places, including balconies or terraces).
* Speak and understand Catalan or Spanish.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete smoke-free rule at home | 3 and 6 months post-baseline
  At recruitment, none of the participants will have a smoke-free home. The primary outcome measure of this study is the number of participants who establish a smoke-free home, meaning those who report that the current home smoking rule is not to smoke anywhere indoors or outdoors (balconies) the home. This will be assessed through a telephone survey using the question: "Which statement best describes the smoking rules in your home?", with response options: 1) Smoking is never allowed in any part of the home, including indoor and outdoor areas such as a balcony or terrace. 2) Smoking is allowed only sometimes or in specific areas within the home. 3) Smoking is allowed anywhere and at any time in the home, meaning there are no smoking restrictions. Participants who select response number one will be considered to have a smoke-free home.

SECONDARY OUTCOMES:
Home smoking frequency | 3 and 6 months post-baseline
  Self-reported outcome. "How often does someone smoke in your home? daily, weekly, monthly, less than monthly, never."
Second-hand smoke exposure at home | Past 7 days; 3 and 6 months post-baseline
  Self-reported outcome. Number of days smoking occurred in the home in the past 7 days
Complete smoke-free vehicle rule | 3 and 6 months post-baseline
  Self-reported outcome. Question: "Which statement best describes the rules about smoking in your car: 1) we do not own a car; 2) there is no norm about smoking in a car and smoking is allowed; 3) smoking is allowed sometimes; 4) smoking is never allowed in a car".
Among participants who smoke: Cigarette consumption | Past 7 days; assessed at 3 and 6 months post-baseline
  Cigarettes smoked per day; days smoked
Among participants who smoke: Cessation attempts | Past 3 months; assessed at 3 and 6 months post-baseline
  Self-reported outcome. Number of quit attempts in the past 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Esteve Fernández, MD, PhD, Principal Investigator — Catalan Insititute of Oncology
Locations (1):
- Catalan Institute of Oncology, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No